CLINICAL TRIAL: NCT05490550
Title: Comparing Insomnia Care As Usual to Digital Augmentation
Brief Title: Comparing Insomnia Care As Usual to Digital Augmentation (CICADA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noctem, LLC (Industry)
Responsible Party: Principal Investigator, Anne Germain, NOCTEM Founder & CEO, Noctem, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JW210372
Record Dates: First submitted 2022-07-30; First posted 2022-08-05 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Chronic Insomnia
Keywords: Insomnia; Cognitive Behavioral Therapy for Insomnia (CBTI); Digital Technology; Adherence Monitoring
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two study arms (COAST-enhanced CBTI or insomnia care as usual) at the site level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COAST-enhanced CBTI (Active Comparator): Patients randomized to COAST will receive CBTI via the COAST platform, with the assistance of a licensed clinician via NOCTEM's digital sleep hub. Participants will utilize the COAST patient app on their smartphone for engagement in insomnia treatment and receipt of clinician's recommendations. COAST clinicians will utilize the COAST web-based portal for adherence monitoring, progress review, and for providing personalized insomnia treatment recommendations.
  Interventions: Behavioral: COAST-enhanced CBTI
- Military Treatment Facility Insomnia Care As Usual (Active Comparator): Patients randomized to the ICAU arm will receive insomnia care as usual by a certified clinician at their respective site, according to current referral and treatment practices.
  Interventions: Behavioral: Military Treatment Facility Insomnia Care As Usual

INTERVENTIONS:
Behavioral: COAST-enhanced CBTI — Participants will receive CBTI delivered through the COAST platform by one of NOCTEM's certified and licensed COAST clinician. Communication between the participant and licensed clinician will occur primarily through COAST's HIPAA-compliant text messaging, but clinicians and patients may elect to connect via telephone calls or HIPAA-compliant secure videoconference if needed.
  Arms: COAST-enhanced CBTI
Behavioral: Military Treatment Facility Insomnia Care As Usual — Participants will receive the insomnia care offered at their site following current delivery practices (i.e., face-to-face or virtual; individual or group format). During the treatment phase, participants randomized to ICAU will be instructed to communicate with their clinicians as needed, according to standard procedures in place.
  Arms: Military Treatment Facility Insomnia Care As Usual

SUMMARY:
The purpose of this pragmatic non-inferiority randomized clinical trial is to evaluate whether Cognitive Behavioral Treatment of Insomnia (CBTI) delivered through a clinical decision support digital platform is non-inferior to insomnia care delivered as usual at three military treatment facilities for treatment of insomnia, symptoms of depression and anxiety, and treatment satisfaction.

DETAILED DESCRIPTION:
Chronic insomnia is pervasive among service members and adversely affects health and readiness. Insomnia rarely remits spontaneously, and sleep-focused treatments are required to reduce or eliminate insomnia. Cognitive Behavioral Treatment of Insomnia (CBTI) is the first line treatment for insomnia. CBTI remains underutilized and is often unavailable in care settings where service members receive sleep healthcare. Digital health technology is one of the strategic components identified by the DHA to support behavioral health, including sleep health. NOCTEM® has developed and validated its Clinician Operated Assistive Sleep Technology (COAST™) platform to scale delivery and access to CBTI. This non-inferiority trial will evaluate and compare the changes in insomnia severity following COAST-enhanced CBTI or insomnia care as usual (ICAU) pre- to post-treatment and at the 3-month follow up. Secondary outcomes of interest include changes in depression and anxiety over time, and patient satisfaction with insomnia care following COAST-enhanced CBTI or ICAU.

ELIGIBILITY:
Inclusion Criteria:

* Active duty service members, men and women, diagnosed with chronic insomnia and deemed eligible for CBTI by their treating clinician.
* Age 18 or older.
* Absence of, or stable, psychiatric, or medical comorbidity(ies), such that they do not compromise safety when completing study procedures.
* If using prescribed sleep medication(s), have received the medication(s) at a stable dosage for at least 4 weeks, with no scheduled change in medication or dosage over the acute intervention phase (up to 12 weeks)
* Owning or ability to use a smartphone (iPhone or Android) that is no older than 5 years old (e.g., iPhone 6, and Android phone with Lollipop 5.0 mobile operating system)

Exclusion Criteria:

* Presence of an untreated or under-treated comorbid sleep disorder that requires independent treatment or that may be exacerbated by sleep restriction or stimuli control, e.g., obstructive sleep apnea (OSA) or rapid-eye-movement (REM) behavior disorder or sleep walking with a history of injury to self or others.
* Acute psychiatric distress associated with marked impairments in functioning or that limits engagement in CBTI, adversely impacts the risk/benefit ratio of participating in the study, or requires immediate attention, as indicated by, but not limited to, the examples listed below. Please note that each referring clinician will determine whether a patient is eligible for the study.
* Having planned or attempted suicide or the harming of others in the past 6 months.
* Seeking and/or receiving treatment at psychiatric clinic facility at a level that requires inpatient or partial hospitalization level of psychiatric care.
* Currently requiring the support of an assigned case manager for services such as coordination of medications, appointments, transportation, and/or for completing activities of daily living.
* Active substance use disorder.
* Past or current psychotic or bipolar disorder or sub-threshold symptoms of psychotic or bipolar disorders.
* Currently pregnant, breastfeeding, or being the parent of a newborn < 3 months old.
* Untreated seizure disorder.
* Suspected, diagnosed, or inadequately treated sleep apnea (less than 4 hours of CPAP use per night).
* Anticipates relocating/moving out of state in the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity | baseline
  Insomnia Severity Index (ISI)
Insomnia Severity | 6-8 week check-in
  Insomnia Severity Index (ISI)
Insomnia Severity | 3-month follow up
  Insomnia Severity Index (ISI)
Symptoms of Depression | baseline
  Patient Health Questionnaire-2 (PHQ-2)
Symptoms of Depression | 6-8 week check-in
  Patient Health Questionnaire-2 (PHQ-2)
Symptoms of Depression | 3-month follow up
  Patient Health Questionnaire-2 (PHQ-2)
Symptoms of Anxiety | baseline
  Generalized Anxiety Disorder 2-item (GAD-2)
Symptoms of Anxiety | 6-8 week check-in
  Generalized Anxiety Disorder 2-item (GAD-2)
Symptoms of Anxiety | 3-month follow up
  Generalized Anxiety Disorder 2-item (GAD-2)
Acceptability of Insomnia Care | 6-8 week check-in
  An adapted version of the Insomnia Treatment Acceptability Scale (ITAS) with ratings of perceived acceptability and treatment preference for both COAST-enhanced CBTI and insomnia care as usual (ICAU).
Satisfaction with Insomnia Care | 6-8 week check in
  Client Satisfaction Questionnaire assessing perceived quality of care, services, and clinicians encountered during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Germain, Principal Investigator — Noctem, LLC
Locations (1):
- Madigan Army Medical Center, Lakewood, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edinger JD, Arnedt JT, Bertisch SM, Carney CE, Harrington JJ, Lichstein KL, Sateia MJ, Troxel WM, Zhou ES, Kazmi U, Heald JL, Martin JL. Behavioral and psychological treatments for chronic insomnia disorder in adults: an American Academy of Sleep Medicine clinical practice guideline. J Clin Sleep Med. 2021 Feb 1;17(2):255-262. doi: 10.5664/jcsm.8986. PMID 33164742
- [Background] Pulantara IW, Parmanto B, Germain A. Clinical Feasibility of a Just-in-Time Adaptive Intervention App (iREST) as a Behavioral Sleep Treatment in a Military Population: Feasibility Comparative Effectiveness Study. J Med Internet Res. 2018 Dec 7;20(12):e10124. doi: 10.2196/10124. PMID 30530452
- [Derived] Germain A, Wolfson M, Brock MS, O'Reilly B, Hearn H, Knowles S, Mysliwiec V, Wallace ML. Digital CBTI hubs as a treatment augmentation strategy in military clinics: study protocol for a pragmatic randomized clinical trial. Trials. 2023 Oct 6;24(1):648. doi: 10.1186/s13063-023-07686-2. PMID 37803393